CLINICAL TRIAL: NCT00307736
Title: A Phase I/II Study of Bevacizumab, Erlotinib and 5-fluorouracil With Concurrent External Beam Radiation Therapy in Locally Advanced Rectal Cancer
Brief Title: Bevacizumab, Erlotinib and 5-Fluorouracil With External Beam Radiation Therapy in Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Dana-Farber Cancer Institute (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Lawrence S. Blaszkowsky, MD, Assistant Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-345
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Rectal Cancer; Adenocarcinoma of the Rectum
Keywords: Fluorouracil; bevacizumab; erlotinib; external beam radiation therapy; EBRT
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy and radiation (Experimental): Continuous infusion 5-fluorouracil 225 mg/M2/d, bevacizumab 5 mg/kg IV q 14 days, erlotinib 50-150 mg orally daily for duration of radiation.
  Interventions: Drug: 5-fluorouracil; Drug: bevacizumab; Drug: erlotinib; Procedure: External beam radiation therapy (EBRT)

INTERVENTIONS:
Drug: 5-fluorouracil — Given as a 24-hour infusion on days 1-14 of each 14-day cycle for a total of 3 cycles.
Drug: bevacizumab — Given intravenously on day 1 of each 14-day cycle for a total of 3 cycles.
Drug: erlotinib — Taken orally on days 1-14 of each 14-day cycle for a total of 3 cycles.
Procedure: External beam radiation therapy (EBRT) — Given on days 1-5 and 8-12

SUMMARY:
The purpose of this study is determine the safety of 5-fluorouracil, bevacizumab and erlotinib when administered in combination with external beam radiation therapy(Phase I portion) as well as to begin to collect information about whether this combination treatment is effective in treating(Phase II portion) patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
* All participants will receive the following drugs: 5-fluorouracil (5-FU) given as a continuous 24-hour infusion; Bevacizumab given intravenously; erlotinib given orally at home. In the Phase I portion, we are looking for the highest dose of erlotinib that can be given safely in combination with the 5-FU, bevacizumab and radiation therapy. Therefore the dose of erlotinib may not be the same for each participant. The dose will increase until we find the highest dose without causing serious or unmanageable side effects.
* Study treatment is given as an outpatient and consists of 14 day cycles with a total of 3 cycles. Patients will be given all three study drugs and radiation therapy on a monday (unless a monday falls on on a holiday). This will be day 1 of the first treatment cycle. 5-FU is given continuously days 1-14. Bevacizumab is given on day 1. Erlotinib will be given on days 1-14. Radiation therapy will be performed on Days 1-5 and 8-12.
* The following tests and procedures will be performed weekly while participants are receiving study treatment: physical examination, measurement of vital signs, height and weight; performance status; blood work, urine sample.
* At the end of treatment the following tests will be performed: physical examination and measurement of vital signs; performance status; blood work; CT scans of chest, abdomen and pelvis. Patients will also be evaluated for surgery at this time. Patients will be followed every three months for the first three years after surgery, then every 6 months for the next two years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary adenocarcinoma of the rectum that begins within 15cm of the anal verge as determined by sigmoidoscopy or colonoscopy
* Clinical T3 or T4 tumors as determined by endoscopic ultrasound and/or rectal MRI
* ECOG performance status of 0-2
* 18 years of age or older
* Creatinine of < 2.0
* Adequate hepatic function
* Adequate hematopoietic function
* Use of effective means of contraception in subjects of child-bearing potential

Exclusion Criteria:

* Evidence of metastatic disease as determined by chest/abdominal/pelvic CT or physical exam
* Prior chemotherapy or radiation therapy for treatment of colorectal cancer
* Prior treatment with 5-FU
* Prior treatment with a tyrosine kinase inhibitor, EGFR inhibitor, or VEGF inhibitor
* Patients must not be receiving any other investigational agent
* Prior malignancy within the last 5 years except for completely excised skin cancer, in situ cervical cancer
* Warfarin anticoagulation
* Co-existent malignant disease
* Current or recent participation in a clinical trial (within 4 weeks from the first day of treatment)
* Pregnancy
* Blood pressure of >150/100 mmHg
* Unstable angina
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant trauma injury within 28 days prior to day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to day 0
* Pregnant or lactating
* Urine protein:creatinine ratio > or equal to one at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to day 0]
* Serious, non-healing wound, ulcer, or bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-05; Primary Completion 2010-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S. Blaszkowsky, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Blaszkowsky LS, Ryan DP, Szymonifka J, Borger DR, Zhu AX, Clark JW, Kwak EL, Mamon HJ, Allen JN, Vasudev E, Shellito PC, Cusack JC, Berger DL, Hong TS. Phase I/II study of neoadjuvant bevacizumab, erlotinib and 5-fluorouracil with concurrent external beam radiation therapy in locally advanced rectal cancer. Ann Oncol. 2014 Jan;25(1):121-6. doi: 10.1093/annonc/mdt516. PMID 24356623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a single center (institutions comprising Dana Farber Partners/Harvard Cancer Center) trial. Subjects were selected upon referral to the respective clinics of the investigators' institution. Patients Patients were enrolled on to the study between May 2006 and December 2009.
Groups:
- Phase 1 (Erlotinib 50mg); Phase 1 (100mg Erlotinib); Phase 1 (150mg Erlotinib); Phase II (100mg Erlotinib): Continuous infusion 5-fluorouracil 225 mg/M2/d, bevacizumab 5 mg/kg IV q 14 days, erlotinib 50-150 mg orally daily for duration of radiation.
  5-fluorouracil: Given as a 24-hour infusion on days 1-14 of each 14-day cycle for a total of 3 cycles.
  bevacizumab: Given intravenously on day 1 of each 14-day cycle for a total of 3 cycles.
  erlotinib: Taken orally on days 1-14 of each 14-day cycle for a total of 3 cycles.
  External beam radiation therapy (EBRT): Given on days 1-5 and 8-12
Period: Overall Study
Arm/Group | Phase 1 (Erlotinib 50mg) | Phase 1 (100mg Erlotinib) | Phase 1 (150mg Erlotinib) | Phase II (100mg Erlotinib)
Started | 3 | 3 | 3 | 23
Completed | 3 | 3 | 0 | 20
Not Completed | 0 | 0 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- 5-fluorocuracil, Bevacizumab, Erlotinib and Radiation: All patients receive chemoradiation with continuous infusion 5-fluorouracil, bevacizumab and erlotinib.
Arm/Group | 5-fluorocuracil, Bevacizumab, Erlotinib and Radiation
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [35 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29
  Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 32
Stage Grouping [Count of Participants; unit: Participants] — The cancer is referred to as Stage II rectal cancer if the pathology report shows that the cancer has penetrated the wall of the rectum, but does not invade any of the local lymph nodes and cannot be detected in other locations in the body The cancer is referred to as Stage III rectal cancer if the pathology report shows that the cancer has invaded any of the local lymph nodes, but cannot be detected in other locations in the body.
  Participants
    II | 11
    III | 21
Clinical staging [Count of Participants; unit: Participants] — MRI or ultrasound determined T stage. Clinical staging is based off of TNM staging (Tumor, Node, Metastasis). The "T" and the following number (0 to 4) are used to describe how deeply the primary tumor has grown into the bowel lining (Tx: primary tumor cannot be evaluated, Tis: refers to carcinoma in situ). The "N" stands for lymph nodes: (Nx: regional lymph nodes cannot be evaluated; N0: no spread to regional lymph nodes; N1: tumor cells found in 1-3 regional lymph nodes; N2: tumor cells found in 4-7 regional lymph nodes). M0: the disease has not spread to a distant part of the body.
  Participants
    T3N0 | 6
    T3N1 | 15
    T3N2M0 | 4
    T3Nx | 4
    T4N0 | 2
    T4N1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Erlotinib When Administered in Combination With 5-fluorouracil (5-FU), Bevacizumab, and External Beam Radiation Therapy
Description: MTD of Erlotinib was determined using a traditional 3 + 3 dose escalation scheme of three dose levels (50,100,150mg). Successive cohorts of 3-6 patients were enrolled into dose escalation cohorts for 14 day cycles. MTD reflects the highest dose of Erlotinib that had ≤1 out of 6 patients with Dose-Limiting Toxicity (DLT) at the highest dose level below the maximally administered dose. The maximally administered dose is the first dose that causes DLT in >33% of patients. DLT was defined as: Any grade 4 neutropenia, Any grade 3 thrombocytopenia, or Any ≥ grade 3 non-hematologic toxicity that results in greater than 7 days interruption in therapy.
Time Frame: 3 years
Measure: Number; unit: mg
Groups:
- 5-FU, Bevacizumab, Erlotinib and Radiation: All patients received chemoradiation with continuous infusion 5-fluorouracil, bevacizumab and erlotinib. (phase 1 participants)
Arm/Group | 5-FU, Bevacizumab, Erlotinib and Radiation
Number analyzed (Participants) | 9
mg | 100

2. Secondary Outcome: Summary of Grade 3 or Greater Toxicity
Description: Summary of grade 3 or greater toxicity by grade and type. All adverse events were evaluated using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
  Grade 3: Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
Time Frame: 3 years
Population: Toxicity was grouped together for all phase I dose cohorts and the phase II cohort in order to summarize all the grade 3 or greater toxicities associated with the combined study therapy, instead of focusing on the dose limiting toxicities from the phase 1 dose escalation of Erlotinib. Grade 3 or higher AE data is not available by dose cohort.
Measure: Number; unit: participants
Groups:
- Grade 3; Grade 4: Continuous infusion 5-fluorouracil 225 mg/M2/d, bevacizumab 5 mg/kg IV q 14 days, erlotinib 50-150 mg orally daily for duration of radiation.
  5-fluorouracil: Given as a 24-hour infusion on days 1-14 of each 14-day cycle for a total of 3 cycles.
  bevacizumab: Given intravenously on day 1 of each 14-day cycle for a total of 3 cycles.
  erlotinib: Taken orally on days 1-14 of each 14-day cycle for a total of 3 cycles.
  External beam radiation therapy (EBRT): Given on days 1-5 and 8-12
Arm/Group | Grade 3 | Grade 4
Number analyzed (Participants) | 32 | 32
participants
  Lymphopenia | 16 | 5
  Diarrhea w/o prior colostomy | 6 | 0
  Hypophosphatemia | 3 | 0
  Rash: acne/acneiform | 2 | 0
  ALT-SGPT | 1 | 0
  AST-SGOT | 1 | 0
  Cardiac-ischemia | 1 | 0
  Colitis | 1 | 0
  Dehydration | 1 | 0
  Fatigue | 1 | 0
  Febrile neutropenia | 0 | 1
  Hypertension | 1 | 0
  Hyperuricemia | 0 | 1
  Hypokalemia | 1 | 0
  Hyponatremia | 1 | 0
  Muco/stomatitis (symptom) oral cavity | 1 | 0
  Muco/stomatitis by exam-oral cavity | 1 | 0
  Proteinuria | 1 | 0
  Radiation dermatitis | 1 | 0
  Rash/desquamation | 1 | 0
  Rectum-pain | 1 | 0

3. Secondary Outcome: Percentage of Participants With Disease-free Survival
Description: Summary of disease free survival at 1, 2, and 3 years. Disease free survival is the length of time after primary treatment for cancer ends that the participant survives without any clinical signs or symptoms of that cancer. The data is shown of the percentage of participants still in disease free survival at one, two, and three years.
Time Frame: 1, 2, 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 5-fluorocuracil, Bevacizumab, Erlotinib and Radiation: Continuous infusion 5-fluorouracil 225 mg/M2/d, bevacizumab 5 mg/kg IV q 14 days, erlotinib 50-150 mg orally daily for duration of radiation.
  5-fluorouracil: Given as a 24-hour infusion on days 1-14 of each 14-day cycle for a total of 3 cycles.
  bevacizumab: Given intravenously on day 1 of each 14-day cycle for a total of 3 cycles.
  erlotinib: Taken orally on days 1-14 of each 14-day cycle for a total of 3 cycles.
  External beam radiation therapy (EBRT): Given on days 1-5 and 8-12
Arm/Group | 5-fluorocuracil, Bevacizumab, Erlotinib and Radiation
Number analyzed (Participants) | 32
percentage of participants
  1 Year | 93.4 [76.2 to 98.3]
  2 Years | 83.4 [64.7 to 92.7]
  3 Years | 75.5 [55.1 to 87.6]

4. Secondary Outcome: Post-operative Complications After Resection of Rectal Cancers Following Preoperative 5-FU, Bevacizumab, Erlotinib, and External Beam Radiation Therapy.
Description: Surgical morbidity following R0 resection with one of the following procedures: abdominal perineal resection, low anterior resection, and low anterior resection with coloanal anastomosis.
Time Frame: 3 years
Population: Total study population excluding one patient who refused surgery.
Measure: Number; unit: participants
Groups:
- Surgery, 5-fluorocuracil, Bevacizumab, Erlotinib and Radiation: Patients undergoing R0 resection following chemotherapy and radiation.
  Continuous infusion 5-fluorouracil 225 mg/M2/d, bevacizumab 5 mg/kg IV q 14 days, erlotinib 50-150 mg orally daily for duration of radiation.
  5-fluorouracil: Given as a 24-hour infusion on days 1-14 of each 14-day cycle for a total of 3 cycles.
  bevacizumab: Given intravenously on day 1 of each 14-day cycle for a total of 3 cycles.
  erlotinib: Taken orally on days 1-14 of each 14-day cycle for a total of 3 cycles.
  External beam radiation therapy (EBRT): Given on days 1-5 and 8-12
Arm/Group | Surgery, 5-fluorocuracil, Bevacizumab, Erlotinib and Radiation
Number analyzed (Participants) | 31
participants
  anastomotic leaks | 4
  intra-abdominal infection | 2
  wound infections | 2
  pulmonary embolus | 1
  small bowel obstruction | 1
  urinary obstruction/retention | 5
  fever | 1

5. Other Pre Specified Outcome: Pathologic Complete Response
Description: The number of subjects who achieved a pathologic complete response as determine by pathologist, following completion of the study therapy. Pathologic complete response represents the absence of residual invasive disease in the rectum and in the regional lymph nodes.
Time Frame: 3 years
Population: Patients who completed study therapy.
Measure: Count of Participants; unit: Participants
Groups:
- Completed Study Therapy: Patients who had pathologic complete response following completion of study therapy.
  All patients receive chemo-radiation with continuous infusion 5-fluorouracil, bevacizumab and erlotinib.
- Underwent Resection: Patients who underwent R0 resection following study therapy
  All patients receive chemoradiation with continuous infusion 5-fluorouracil, bevacizumab and erlotinib.
- Treated at MTD: Patients who were treated with erlotinib at maximum tolerated dose, along with standard study therapy.
  All patients receive chemoradiation with continuous infusion of 5-fluorouracil, bevacizumab and erlotinib.
Arm/Group | Completed Study Therapy | Underwent Resection | Treated at MTD
Number analyzed (Participants) | 27 | 31 | 26
Participants | 9 | 10 | 7

ADVERSE EVENTS:
Time Frame: 3 years
Description: Patients were evaluated for adverse events at each study visit for the duration of their participation in the study. Safety evaluations consisted of medical interviews, recording of adverse events, physical examinations, blood pressure, and laboratory measurements. Patients discontinued from the treatment phase of the study for any reason would be evaluated ~30 days. Adverse event data was aggregated for phase 1 and 2 portion of the study. Adverse event data by dose cohort is not available.
Arm/Group | 5-fluorocuracil, Bevacizumab, Erlotinib and Radiation
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 8/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-fluorocuracil, Bevacizumab, Erlotinib and Radiation (N=32)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Cardiac Ischemia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-fluorocuracil, Bevacizumab, Erlotinib and Radiation (N=32)
Abdomen pain (Gastrointestinal disorders) | 12 (19)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (6)
Allergic reaction (Immune system disorders) | 3 (3)
Allergic rhinitis (Immune system disorders) | 2 (2)
ALT- SGPT (Metabolism and nutrition disorders) | 8 (10)
Anorexia (Gastrointestinal disorders) | 16 (28)
Anus- pain (Gastrointestinal disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
AST- SGOT (Metabolism and nutrition disorders) | 10 (13)
Back- pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bicarbonate (Metabolism and nutrition disorders) | 2 (3)
Bilirubin (Metabolism and nutrition disorders) | 5 (9)
Confusion (Nervous system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Creatinine (Metabolism and nutrition disorders) | 2 (2)
Cystitis (Renal and urinary disorders) | 2 (3)
Dehydration (Gastrointestinal disorders) | 7 (9)
Depression (Psychiatric disorders) | 2 (3)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 29 (65)
Dizziness (Nervous system disorders) | 5 (8)
Dry mouth (Gastrointestinal disorders) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (6)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Extremity-limb- pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Fatigue (General disorders) | 29 (67)
Fever w/o neutropenia (General disorders) | 3 (6)
Flatulence (Gastrointestinal disorders) | 4 (8)
Flushing (Skin and subcutaneous tissue disorders) | 2 (3)
GI-other (Gastrointestinal disorders) | 6 (10)
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 4 (5)
Head/headache (Nervous system disorders) | 6 (7)
Hemoglobin (Blood and lymphatic system disorders) | 12 (22)
Hemorrhage-other (Blood and lymphatic system disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 7 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (28)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Cardiac disorders) | 3 (4)
Hypoalbuminemia (Blood and lymphatic system disorders) | 7 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 13 (16)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5)
Insomnia (General disorders) | 8 (15)
Leukocytes (Blood and lymphatic system disorders) | 15 (26)
Lymphopenia (Blood and lymphatic system disorders) | 29 (73)
Memory impairment (Nervous system disorders) | 2 (4)
Mucositis/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 11 (23)
Mucositis/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 8 (13)
Muscle- pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 24 (41)
Neuropathy-sensory (Nervous system disorders) | 3 (4)
Neutrophils (Blood and lymphatic system disorders) | 2 (3)
Nose- hemorrhage (Respiratory, thoracic and mediastinal disorders) | 9 (14)
Oral cavity- pain (Gastrointestinal disorders) | 2 (3)
Oral gums- pain (Gastrointestinal disorders) | 2 (2)
Pain-other (General disorders) | 2 (3)
Pelvic- pain (Reproductive system and breast disorders) | 3 (5)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Proctitis (Reproductive system and breast disorders) | 2 (2)
Proteinuria (Metabolism and nutrition disorders) | 6 (9)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5 (7)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 10 (15)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (15)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 23 (59)
Rectum- hemorrhage (Gastrointestinal disorders) | 13 (21)
Rectum- pain (Gastrointestinal disorders) | 24 (38)
Renal/GU-other (Renal and urinary disorders) | 2 (2)
Rigors/chills (General disorders) | 7 (8)
Skin-other (Skin and subcutaneous tissue disorders) | 8 (12)
Sweating (General disorders) | 2 (2)
Taste disturbance (Gastrointestinal disorders) | 4 (5)
Throat/pharynx/larynx- pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Urinary frequency/urgency (Renal and urinary disorders) | 6 (12)
Urinary retention (Renal and urinary disorders) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3)
Vagina- pain (Reproductive system and breast disorders) | 2 (4)
Vision-blurred (Eye disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)
Weight loss (General disorders) | 14 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No